CLINICAL TRIAL: NCT00946660
Title: Human Laboratory Model of Cocaine Treatment: Behavioral Economic Analysis: Study 1
Brief Title: Non-Treatment Study of Factors Affecting Cocaine Drug Choice
Acronym: CTA
Status: Completed | Type: Observational
Sponsor: Wayne State University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Mark Greenwald, PhD, Principal Investigator, Wayne State University
Other Study IDs: NIDA-DA026861; R01DA026861 (NIH); DCNBR
Record Dates: First submitted 2009-07-24; First posted 2009-07-27 (Estimated); Last update posted 2012-06-05 (Estimated); Status verified 2012-06

CONDITIONS: Cocaine Abuse or Dependence; Cocaine Related Disorders
Keywords: Contingency Management; Drug Self-Administration
MeSH Terms: conditions — Cocaine-Related Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole Blood
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This research deals with behaviors that are part of drug dependence. The purpose is to study how certain factors, including money, the amount of drug available, and the amount of work effort, affect cocaine drug choice. Specifically, we will examine the effects of two issues/factors. The first is how hard individuals are willing to work to obtain a drug; the second is how much drug would individuals choose instead of money, when the amount of probability of money is predictable or unpredictable.

DETAILED DESCRIPTION:
Outpatient Phase: Participants will be outpatients and must come to the Jefferson Avenue Research Program three times a week (Mon-Wed-Fri). This phase will last two weeks. At each visit participants will be asked to provide a urine sample and to complete questionnaires that ask about substance use.

Inpatient Phase: Participants will live on an inpatient research unit at least 2 consecutive nights and possibly up to 20 consecutive nights. Participants cannot have visitors and will not be allowed to leave the inpatient unit (except with a staff escort) unless they drop out of the study. We will collect daily urine samples to make sure participants are not using any drugs except those in the study.

Participants will take part in multiple trials (up to 11 experimental sessions) where they will be given a standard amount of powder (identified as Drug A or Drug B) to inhale through a straw into their nose. The powder will contain placebo (a powder containing no drug) or different doses of cocaine. We will measure how participants are feeling using questionnaires and we will record vital signs-including breathing rate, blood oxygen level, heart rate, and blood pressure.

Participants will also be asked to perform a 3-hour computer task that allows them to work for Drug A, Drug B, or money. At the end of the computer task participants will receive the amount of drug they earned and a receipt for the amount of money they earned.

To complete the study, a minimum stay of 16 inpatient nights is required. The maximum stay is 20 inpatient nights.

ELIGIBILITY:
Inclusion Criteria:

* Male or female volunteers(18-55 years of age).
* Must meet criteria for Cocaine Abuse or Dependence and wish to participate in research.
* Positive urine test for cocaine.
* Candidates must be in good health to be eligible.
* All candidates must receive routine medical (history and physical) exam with standard laboratory tests (complete blood chemistry, urinalysis, urine pregnancy test for females, tuberculin screening), and 12-lead ECG at the initial screening visit.

Exclusion Criteria:

* Serious psychiatric illness (e.g. psychosis, bipolar, suicide attempts, major depression that is not substance-induced)
* Substance use disorder other than cocaine abuse or dependence, nicotine dependence, alcohol abuse, sedative abuse or marijuana abuse.
* Neurological diseases (e.g. stroke, seizures); cardiovascular problems (e.g. myocardial infarction, angina, systolic BP >160 or <95 mmHg, diastolic BP >95 mmHg, or clinically abnormal ECG); pulmonary diseases (e.g. asthma, TB); systemic diseases (e.g. hepatitis, autoimmune diseases)
* Cognitive impairment
* Exposed in past 30 days to medications that would increase study risk (e.g. toxicity to major organ systems, psychotropics, asthma inhalers, or interactions with study drugs)
* Pregnant (urine HCG), lactating (self-report), or if heterosexually active and not using (self-report) medically approved birth control measures (oral or depot contraceptives, IUD, condom/foam, sterilization, tubal ligation)
* Seeking treatment or being treated for a substance use disorder.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Cocaine abusing or dependent research volunteers
Sampling Method: Non-Probability Sample
Enrollment: 16 (Estimated)
Dates: Start 2009-07; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Greenwald, PhD, Principal Investigator — Wayne State University
Locations (1):
- Wayne State University, Detroit, Michigan, United States

REFERENCES:
- [Derived] Greenwald MK, Ledgerwood DM, Lundahl LH, Steinmiller CL. Effect of experimental analogs of contingency management treatment on cocaine seeking behavior. Drug Alcohol Depend. 2014 Jun 1;139:164-8. doi: 10.1016/j.drugalcdep.2014.03.009. Epub 2014 Mar 19. PMID 24685561